CLINICAL TRIAL: NCT00165386
Title: MRI-guided Bone Marrow Biopsies of Advanced CaP Patients
Brief Title: MRI-guided Bone Marrow Biopsies of Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-108
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Prostate Cancer
Keywords: MRI-guided bone marrow biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging
Procedure: Bone Marrow Biopsy

SUMMARY:
The purpose of this study is to target lesions of the prostate in the bone and to biopsy these lesions using MRI to identify the areas.

DETAILED DESCRIPTION:
* This study involves a one-time, MRI-guided bone marrow biopsy. Prior to this procedure, patients will need to have a bone scan performed within the last three months and a PSA blood test drawn within one month of registration to the study.
* Patients are also required to participate in the DFCI research study "Collection of Specimens and Clinical Data for Patients with Prostate Cancer or at High Risk for Prostate Cancer".

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of prostate cancer
* Bone scan consistent with or suspicious of metastatic prostate cancer within last three months
* Platelet count > 50,000/ul
* PT and aPTT < 1.5 x control
* At least one week removed from taking aspirin or coumadin
* Currently participating in protocol "Collection of Specimens and Clinical Data for Patients with Prostate Cancer or at High Risk for Prostate Cancer"

Exclusion Criteria:

* Devices incompatible to MR studies (e.g. pacemakers, ear implants, etc.)

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2001-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To compare the yield of detecting metastatic prostate cancer tissue using MRI-guided bone marrow needle biopsies to that of historical controls obtained through unguided biopsies.

SECONDARY OUTCOMES:
To evaluate the sensitivity of radiographic bone marrow changes detected by MRI for prostate cancer, as determined by the pathologic findings from bone marrow biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States